CLINICAL TRIAL: NCT06654830
Title: Robotic-assisted Versus Video-assisted Thoracoscopic Thymectomy for Thymic Epithelial Tumor in Stage I-II: a Prospective, Multi-center, Randomized Controlled Trial
Brief Title: RATT Vs. VATT for Early-stage TETs
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Qilu Hospital of Shandong University (Other); The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2024455
Record Dates: First submitted 2024-09-28; First posted 2024-10-23 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Thymic Epithelial Tumor
Keywords: thymic epithelial tumor; robot-assisted; video-assisted; thoracoscopic thymectomy
MeSH Terms: conditions — Thymic epithelial tumor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RATT (Experimental): robotic-assisted thoracoscopic thymectomy
  Interventions: Procedure: RATT
- VATT (Active Comparator): video-assisted thoracoscopic thymectomy
  Interventions: Procedure: VATT

INTERVENTIONS:
Procedure: RATT — Robotic-assisted thoracoscopic thymectomy (RATT) will be performed using Da Vinci Robotic Surgical Systems.
  Arms: RATT
Procedure: VATT — Video-assisted thoracoscopic thymectomy (VATT) was performed using traditional thoracoscopic systems.
  Arms: VATT

SUMMARY:
This study is a prospective, multicenter, phase II randomized controlled trial. We plan to screen 100 eligible thymoma patients for robotic-assisted thoracoscopic thymectomy (RATT) or video-assisted thoracoscopic thymectomy (VATT) at three medical centers in China. The trial was aimed to compare the perioperative outcomes between the two approaches.

ELIGIBILITY:
Inclusion Criteria:

* Thymoma was diagnosed by chest enhanced CT or MRI (clinical stage: Masaoka Koga I-II) with AJCC/UICC TNM grade system (9th edition).

The patients whose tumor diameter was not larger than 8 cm; The patients with the estimated survival time should be over 12 months; ASA grade：1-2; The patients should have no functional disorders in main organs; The patients should be able to understand our research and sign the informed consent.

Exclusion Criteria:

* Imaging examination showed that the tumor had invasion of surrounding organs, pleural or pericardial dissemination, lymphatic or hematogenous metastasis; Patients with myasthenia gravis; Patients had undergone a sternotomy; The patients have proved history of congestive heart failure, angina without good control with medicine; ECG-proved penetrating myocardial infarction; hypertension with bad control; valvulopathy with clinical significance; arrhythmia with high risk and out of control; The patients have severe systematic intercurrent disease, such as active infection or poorly controlled diabetes; coagulation disorders; hemorrhagic tendency or under treatment of thrombolysis or anticoagulant therapy; Female who is positive for serum pregnancy test or during lactation period; The patients have history of organ transplantation (including autologous bone marrow transplantation and peripheral stem cell transplantation; The patients have history of peripheral nerve system disorders, obvious mental disorders or central nerve system disorders; The patients attend other clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative draingage volume | Up to 7 days.
  Postoperative draingage volume is the total draingage volume after surgery.

SECONDARY OUTCOMES:
complete recestion rate | Up to 7 days.
the counts of lymph node sampling | From the time at start of the surgery to the time at end of the surgery. Up to 7 days.
operative time | From the time at start of the surgery to the time at end of the surgery. Up to 7 days.
bleeding volume | From the time at start of the surgery to the time at end of the surgery. Up to 7 days.
duration of drainage | from the day of the surgery to the day of removal of drainage tubes. Up to 7 days.
postoperative hospital stays | from the day of the surgery to the day of discharge. Up to 30 days
re-operation rate | from the day of the surgery to the day of discharge. Up to 7 days
C-reactive protein level at postoperaive day 1 | from the day of the surgery to the day of discharge. Up to 7 days
C-reactive protein level at postoperaive day 2 | from the day of the surgery to the day of discharge. Up to 7 days
serum interleukin-6 level at postoperaive day 1 | from the day of the surgery to the day of discharge. Up to 7 days
serum interleukin-6 level at postoperaive day 2 | from the day of the surgery to the day of discharge. Up to 7 days
serum procalcitonin level at postoperaive day 1 | from the day of the surgery to the day of discharge. Up to 7 days
serum procalcitonin level at postoperaive day 2 | from the day of the surgery to the day of discharge. Up to 7 days
pain visual analogue scale score at postoperative day 1, 2, 3 and 7 | from the day of the surgery to the postoperative day 7. Up to 7 days
quality of life score at postoperative day 30, 60 and 180 | from the day of the surgery to the postoperative day 180. Up to 180 days
complication rate | from the day of the surgery to the day of discharge. Up to 30 days
3-year disease-free survival | from the day of the surgery to the postoperative 3 years. Up to 3 years
3-year overall survival | from the day of the surgery to the postoperative 3 years. Up to 3 years

IPD SHARING:
Plan to Share IPD: No
National policy.

REFERENCES:
- [Derived] Wang S, Zhu J, Sun Z, Jiang J, Wu B, Liang F, Zheng Y, Yang X, Jiang X, Ao YQ, Gao J, Tan L, Qi Y, Yue W, Ding J. Robot-assisted versus video-assisted thoracoscopic thymectomy for stage I-II thymic epithelial tumour: a protocol for the first multicentre, randomised controlled clinical trial. BMJ Open. 2025 May 28;15(5):e095802. doi: 10.1136/bmjopen-2024-095802. PMID 40441770